CLINICAL TRIAL: NCT05159388
Title: A First in Human Phase 1-2 Open-Label, Multicenter, Dose Escalation and Expansion Study of PRS-344/S095012 in Patients With Solid Tumors
Brief Title: A Study of PRS-344/S095012 (PD-L1x4-1BB Bispecific Antibody-Anticalin Fusion) in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95012-001; 2019-003456-36 (EudraCT Number)
Record Dates: First submitted 2021-11-15; First posted 2021-12-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
Keywords: Solid Tumor = Phase 1/2; Open-label; Dose escalation; Metastatic; PRS-344; S095012; PRS-344/S095012; Anticalin protein; Bi-specific; 4-1BB; CD137; PD-L1
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRS-344/S095012 (Experimental): PRS-344/S095012
  Interventions: Drug: PRS-344/S095012

INTERVENTIONS:
Drug: PRS-344/S095012 — PRS-344/S095012 Monotherapy

SUMMARY:
This is a first-in-human (FIH), phase 1/2, multi center, open-label, dose escalation and cohort expansion study designed to determine the safety and tolerability of PRS-344/S095012 in patients with advanced and/or metastatic solid tumors.

DETAILED DESCRIPTION:
The trial is an open-label, multi-center safety trial of PRS-344/S095012. The trial consists of two parts, a dose escalation part (phase 1, first-in-human (FIH) and an expansion part (phase 2)). The expansion part of the trial will be initiated once the optimal biological dose (OBD) has been determined.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years on the day the consent is signed.
2. Patients with histologically confirmed diagnosis of unresectable, locally advanced or metastatic solid tumor for which standard treatment options are not available, no longer effective, or not tolerated.
3. Patient should have a documented disease progression on prior therapy before entry into this study.
4. Patients must have at least one measurable target lesion as per RECIST 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Patient with no available archived material must have one or more tumor lesions amenable to biopsy.
7. Adequate organ function as assessed by laboratory tests within 7 days prior to pretreatment with obinutuzumab.
8. A female patient must use a highly effective method of birth control during study treatment and for 120 days after last dose of PRS-344/S095012, or 18 months after the last obinutuzumab infusion, whichever comes the latest.

Exclusion Criteria:

1. Patients with previously treated brain metastases may participate provided they are radiologically stable, clinically asymptomatic and are off immunosuppressive therapies for at least 4 weeks. Low dose of steroid <10 mg/day prednisone or equivalent) is allowed.
2. Patients who have received prior:

   1. Small molecule inhibitors, and/or other similar investigational agent: ≤ 2 weeks or 5 half-lives, whichever is shorter.
   2. Chemotherapy, other monoclonal antibodies, antibody-drug conjugates, or other similar experimental therapies: ≤3 weeks or 5 half-lives, whichever is shorter.
   3. Radioimmunoconjugates or other similar experimental therapies ≤6 weeks or 5 half-lives, whichever is shorter.
3. Patients who have received 4-1BB agonists in the past.
4. Patients who had a major surgery within 4 weeks prior to first administration of IMP.
5. History of progressive multifocal leukoencephalopathy.
6. Active tuberculosis requiring treatment within 3 years prior to the start of treatment or a suspicion of latent tuberculosis by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Safety measurements | 28 days
  Phase 1: Incidence of dose-limiting toxicities (DLTs) over the first 28-days of study treatment
Safety Measurements | time on trial, average of 6 months
  Phase 1: Incidence of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Safety Measurements | time on trial, average of 6 months
  Phase 1: Discontinuation of study treatment due to an AE
Objective Response (OR) | Through study completion up to 24 months
  Phase 2: Defined as Complete Response (CR) plus Partial Response (PR). For arms 1 and 2, per central assessment according to RECIST v1.1 criteria. For Arm 3, per central assessment and composite response criteria (digital medical photography and/or imaging as per RECIST v1.1)

SECONDARY OUTCOMES:
Mean PRS-344/S095012 concentrations at the end of the infusion | Through study completion up to 24 months
  Phase 1
Mean PRS-344/S095012 trough concentrations (Ctrough) | Through study completion up to 24 months
  Phase 1
Detection of anti-drug antibodies (ADA) against PRS-344/S095012 | Through study completion up to 24 months
  Phase 1 and 2
Objective Response (OR) | Through study completion up to 24 months
  Phase 1 and 2: Defined as Complete Response (CR) plus Partial Response (PR), per investigator assessment
Duration of Response (DoR) | Through study completion up to 24 months
  Phase 1 and 2: Defined as the time from first demonstration of response to progression or death, whichever occurs first
Progression-free Survival (PFS) | Through study completion up to 24 months
  Phase 1 and 2: Defined as the time from the first dose of treatment to first documented disease progression or death due to any cause, whichever occurs first
Overall Survival (OS) | Through study completion up to 24 months
  Phase 1 and 2: Defined as the time from first dose of study drug to death due to any cause
Disease Control (DC) | Through study completion up to 24 months
  Phase 2: The proportion of patients who achieved SD, PR, or CR (based on patient's best response)
Time to Response (TTR) | Through study completion up to 24 months
  Phase 2: The time from the first dose of PRS-344/S095012 to the first documentation of CR or PR
Safety measurements | time on trial, average of 6 months
  Phase 2: Incidence of adverse events (AEs)
Safety measurements | time on trial, average of 6 months
  Phase 2: Incidence of serious adverse events (AEs)
Serum concentrations of PRS-344/S095012 | Through study completion up to 24 months
  Phase 2

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Carolina Bio Oncology, Huntersville, North Carolina
  - NEXT Oncology, San Antonio, Texas
- Australia (3):
  - Cabrini Oncology Research, Malvern, Victoria
  - Chris O'Brian Lifehouse, Camperdown
  - The Queen Elizabeth Hospital, Woodville South
- Belgium (3):
  - Institute Jules Bordet, Brussels
  - Universitair Ziekenhuis, Edegem
  - U.Z. Gent Medical Oncology, Ghent
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - START, Madrid
  - Hospital Universitario Gregorio, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jungels C, Kotecki N, Calvo E, Garralda E, Price T, Zahn X, Abbas A, Mahnke L, Rauschning W, Morales-Kastresana A, Lucia Pattarini L, Bossenmaier B, Scholer-Dahirel A, Demuth T, Legrande J. Abstract CT255: Study of PRS-344/S095012 a PD-L1/4-1BB bispecific antibody-Anticalin®-fusion in patients with solid tumors. Canc Res. 2022 Jun 15;82(12_Supplement):CT255. doi: https://doi.org/10.1158/1538-7445.AM2022-CT255